CLINICAL TRIAL: NCT05624827
Title: The Role of FAM19A4 and Hsa-mir-124 Methylation in Predicting Prognosis of Untreated Cervical Intraepithelial Neoplasia 2 (CIN 2)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRP-2021/02-04
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-05

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2; DNA Methylation
Keywords: CIN 2 prognosis; DNA hypermethylation; FAM19A4; hsa-mir-124; tumor suppressor genes; diagnostic implications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with CIN 2 and under 36 years old (Experimental): We will analyze patients under 36 years old (≤ 35) with histological confirmed CIN 2 lesions and without any additional risk factors.
  Interventions: Diagnostic Test: Testing DNA methylation test for predicting prognosis of untreated CIN 2

INTERVENTIONS:
Diagnostic Test: Testing DNA methylation test for predicting prognosis of untreated CIN 2 — After being diagnosed with CIN 2, patients will first be contacted by telephone and invited to participate in the study. If patients agree to participate in the research, they will sign a consent to participate in the research. After that, we will perform a colposcopy and take a cervical swab for analysis with the QIAsure Methylation Test Kit (Qiagen, Gaithersburg, USA), which will determine the methylation of tumor suppressor genes FAM19A4 and has-mir-124. Patients will complete a questionnaire. The total duration of tracking in both groups will be two years. The QIAsure Methylation Test will be performed to analyze methylation. It is a methylation-specific PCR test that detects hypermethylation of the tumor promoter suppressor genes FAM19A4 and has-mir-124. The samples on which we will use this test are bisulfite-converted DNA obtained by triage test for high-risk HPV - Hybrid Capture 2 HPV DNA Test (hc2, Qiagen, Gaithersburg, USA).

SUMMARY:
High-risk precancerous cervical lesions are divided into stage 2 and 3 cervical intraepithelial neoplasia (CIN 2 and 3). CIN 3 represents a direct pre-stage of invasive cancer, has a high rate of progression and a high degree of agreement with the final histological diagnosis. In CIN 2 lesions, the rate of agreement with the final histological diagnosis is lower and the rate of spontaneous regression is higher. Due to the higher rate of regression and possible complications after excisional treatment, conservative active monitoring can be considered in selected young CIN 2 patients. A recent meta-analysis reported a high rate of spontaneous clinical regression of CIN 2, particularly in women under 30 years old. There are currently no prospectively validated prognostic biomarkers to determine which CIN 2 will progress to higher grade and which will regress to lower grade of change. Recent research has studied HPV methylation and microbiome analysis as biomarkers. A number of studies have shown that host cell DNA methylation levels in cervical scrapes increase with underlying cervical disease severity and are highest in cervical cancer. DNA methylation involves the covalent binding of a methyl group to the 5´ position of a cytosine molecule in CpG dinucleotides. Besides global hypomethylation, the overall loss of methylation during carcinogenesis, resulting in chromosomal instability, and the silencing of tumour suppressor genes by local hypermethylation of CpG-rich promoter regions contribute to cancer development. Gene promoter methylation can be easily accessed by sensitive, quantitative methylation-specific PCR providing an objective test outcome. The aim of this study was to determine the effect of the methylation rate of two suppressor genes- FAM19A4 and hsa-mir-124 on the rate of CIN 2 regression, persistence or progression in women younger than 36 years (≤35 years old).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CIN 2 (with biopsy of colposcopically suspicious changes in the cervix)
* Age under 30 years
* Satisfactory colposcopy (transformation zone fully visible)
* Size of change below 75% of transformation zone
* The change in the ectocervix is fully visible
* Age 30-35 years, if the patient is non-smoker and the change in the cervix does not exceed 50% of the area of the transformation zone
* Signing an informed consent to participate in the survey
* Willingness to perform inspections every 6 months

Exclusion Criteria:

* Age 36 years or older
* Unsatisfactory colposcopy (transformation zone not fully visible)
* Size of change exceeds 75% of the transformation zone
* The change in the ectocervix is not completely visible
* Age 30-35 years for smokers or if the change exceeds 50% of the area of the transformation zone
* Suspicted glandular precancerous changes
* Histologically verified CIN 2 with cytological changes of glandular cells
* Colposcopically suspected invasive disease
* Histologically verified CIN 2 and histologically verified AIS
* Histologically verified CIN 2 and histologically verified invasive cancer elsewhere in the cervix
* Refusal to sign participation in the survey
* Unwillingness to perform control examinations
* Weakness of an immune system
* Cervical conization performed in the past
* Treatment with local immunomodulators

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Impact of the degree of methylation on progression of CIN 2 | two years
  The primary clinical outcome will be the effect of the degree of methylation on the progression of CIN 2 to CIN 3+ (CIN 3 and cervical cancer).

SECONDARY OUTCOMES:
Rate of progression of CIN 2 | two years
  The secondary clinical outcome will be the rate of progression of CIN 2 to CIN 3+, the rate of clinical decline to normal histological picture (˂ CIN 1) and the rate of persistence of precancerous change after two years (CIN 2 or persistent CIN 1).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code